CLINICAL TRIAL: NCT03899909
Title: A First-in-human, Randomized, Double-blind, Placebo-controlled, Single Centre Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Single and Multiple Ascending Oral Doses of GLPG3121 for 13 Days in Adult, Healthy, Male Subjects.
Brief Title: A Study to Evaluate the Effects of a Single and Multiple Oral Doses of GLPG3121 in Adult, Healthy, Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Galapagos NV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: GLPG3121-CL-101; 2018-002174-40 (EudraCT Number)
Record Dates: First submitted 2019-04-01; First posted 2019-04-02 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- GLPG3121 SAD (Experimental): Single doses of GLPG3121 at up to 6 dose levels in ascending order
  Interventions: Drug: GLPG3121 SAD
- Placebo SAD (Placebo Comparator): Single doses of placebo
  Interventions: Drug: Placebo SAD
- GLPG3121 MAD (Experimental): Multiple doses of GLPG3121 at up to 4 dose levels in ascending order
  Interventions: Drug: GLPG3121 MAD
- Placebo MAD (Placebo Comparator): Multiple doses of placebo
  Interventions: Drug: Placebo MAD

INTERVENTIONS:
Drug: GLPG3121 SAD — GLPG3121 oral suspension, single ascending doses
  Arms: GLPG3121 SAD
Drug: Placebo SAD — Placebo oral suspension
  Arms: Placebo SAD
Drug: GLPG3121 MAD — GLPG3121 oral suspension, multiple ascending doses, daily for 13 days
  Arms: GLPG3121 MAD
Drug: Placebo MAD — Placebo oral suspension, daily for 13 days
  Arms: Placebo MAD

SUMMARY:
This study is a first-in-human, Phase I, randomized, double-blind, placebo controlled, dose-escalation study to evaluate the safety, tolerability, pharmacokinetics and pharmacodynamics of GLPG3121 after oral single ascending doses (SAD) of GLPG3121 (part 1) and after oral multiple ascending doses (MAD) for 13 days of GLPG3121 (part 2) in healthy male subjects.

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to comply with the protocol requirements and signing the Informed Consent Form (ICF) as approved by the Independent Ethical Committee (IEC)/Institutional Review Board (IRB), prior to any screening evaluations.
* Male between 18 to 55 years of age (extremes included), on the date of signing the ICF.
* A Body Mass Index (BMI) between 18.0 to 30.0 kg/m2, inclusive.
* Judged to be in good health by the investigator based upon the results of a medical history, physical examination, vital signs, (triplicate) 12-lead electrocardiogram (ECG), and fasting clinical laboratory safety tests, available at screening and prior to randomization. Hemoglobin, neutrophil, lymphocyte, and platelet counts must not be below the lower limit of normal range. Bilirubin, aspartate aminotransferase (AST), and alanine aminotransferase (ALT) must be no greater than 1.5x the upper limit of normal range (ULN). Other clinical laboratory safety test results must be within the reference ranges or test results that are outside the reference ranges need to be considered nonclinically significant in the opinion of the investigator.

Exclusion Criteria:

* Known hypersensitivity to investigational medicinal product (IMP) ingredients or history of a significant allergic reaction to IMP ingredients as determined by the investigator.
* Known contraindication or hypersensitivity to interferon-α (IFN-α) or any component of Intron-A® (Note: this criterion is only applicable to subjects in the MAD part).
* Having any illness, judged by the investigator as clinically significant, in the 3 months prior to first dosing of the IMP.
* Presence or sequelae of gastrointestinal, liver, kidney (creatinine clearance ≤80 mL/min using the Cockcroft-Gault formula: if calculated result is ≤80 mL/min a 24-hours urine collection to assess creatinine clearance can be done) or other conditions known to interfere with the absorption, distribution, metabolism, or excretion of drugs.
* History of malignancy within the past 5 years prior to screening with the exception of excised and curatively treated non-metastatic basal cell carcinoma or squamous cell carcinoma of the skin.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2019-03-29 (Actual); Primary Completion 2019-06-03 (Actual); Study Completion 2019-06-03 (Actual)

PRIMARY OUTCOMES:
Frequency and severity of treatment emergent adverse events (TEAEs), treatment-emergent serious adverse events, and TEAEs leading to treatment discontinuations. | From screening through study completion, an average of 6 months.
  To evaluate the safety and tolerability of single and multiple ascending oral doses of GLPG3121, in adult, healthy, male subjects compared with placebo.

SECONDARY OUTCOMES:
Maximum observed plasma concentration (Cmax) of GLPG3121 (μg/mL) | Between Day 1 pre-dose and Day 16
  To evaluate the pharmacokinetics (PK) of single and multiple ascending oral doses of GLPG3121, in adult, healthy, male subjects
Area under curve (AUC) of GLPG3121 (μg.h/mL) | Between Day 1 pre-dose and Day 16
  To evaluate the PK of single and multiple ascending oral doses of GLPG3121, in adult, healthy, male subjects
Terminal elimination half-life (t1/2) of GLPG3121 (h) | Between Day 1 pre-dose and Day 16
  To evaluate the PK of single and multiple ascending oral doses of GLPG3121, in adult, healthy, male subjects

CONTACTS AND LOCATIONS:
Overall Officials: Magdalena Petkova, MD, Study Director — Galapagos NV
Locations (1):
- SGS Belgium NV - Clinical Pharmacology Unit Antwerp, Antwerp, Belgium

IPD SHARING:
Plan to Share IPD: No